CLINICAL TRIAL: NCT00542880
Title: A Double-blind, Randomised, Cross-over, Multi-centre Study, to Evaluate Onset of Effect in the Morning in Patients With Severe Chronic Obstructive Pulmonary Disease (COPD) Treated With Symbicort®Turbuhaler® 320/9 μg, Compared With Seretide® Diskus® 50/500 μg, Both Given as One Inhalation Twice Daily for One Week Each.
Brief Title: Evaluation of Onset of Effect in Patients With Severe Chronic Obstructive Pulmonary Disease (COPD) Treated With Symbicort® Compared to Seretide®
Acronym: SPEED
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: D5892C00016
Record Dates: First submitted 2007-10-10; First posted 2007-10-12 (Estimated); Results first posted 2012-08-30 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-07

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; Symbicort; Seretide
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide, Formoterol Fumarate Drug Combination; Budesonide; Formoterol Fumarate; Salmeterol Xinafoate; Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Symbicort Turbuhaler First, then Seretide Diskus (Experimental): Symbicort Turbuhaler (budesonide/formoterol) 320/9 μg First, then Seretide Diskus (salmeterol/fluticasone) 50/500 μg
  Interventions: Drug: Symbicort Turbuhaler (budesonide/formoterol) 320/9 μg; Drug: Seretide Diskus (salmeterol/fluticasone) 50/500 μg
- Seretide Diskus First, then Symbicort Turbuhaler (Experimental): Seretide Diskus (salmeterol/fluticasone) 50/500 μg First, then Symbicort Turbuhaler (budesonide/formoterol) 320/9 μg
  Interventions: Drug: Symbicort Turbuhaler (budesonide/formoterol) 320/9 μg; Drug: Seretide Diskus (salmeterol/fluticasone) 50/500 μg

INTERVENTIONS:
Drug: Symbicort Turbuhaler (budesonide/formoterol) 320/9 μg
Drug: Seretide Diskus (salmeterol/fluticasone) 50/500 μg

SUMMARY:
This study is to assess the effects with two different inhaled respiratory medications with regards to improvement of lung function, symptoms and morning activities.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient, female or male aged ≥40 years, diagnosis of COPD with symptoms for at least 2 years
* FEV1 ≤50% of predicted normal value, pre-bronchodilator, FEV1/VC <70%
* Pre-bronchodilator

Exclusion Criteria:

* Current respiratory tract disorder other than COPD
* History of asthma or rhinitis
* Significant or unstable cardiovascular disorder

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2007-09; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Andersson, MD, Study Director — AstraZeneca; Martyn R Partridge, MD FRCP, Principal Investigator — Faculty of Medicine, Imperial College, NHLI at Charing Cross Hospital, LONDON, UK
Locations (59):
- Argentina (5):
  - Research Site, Monte Grande, Buenos Aires
  - Research Site, Quilmes, Buenos Aires
  - Research Site, San Miguel de Tucumán, Tucumán Province
  - Research Site, Ciudad Autonoma de Bs. As.
  - Research Site, Ciudad de Buenos Aires
- Australia (7):
  - Research Site, Concord, New South Wales
  - Research Site, Adelaide, South Australia
  - Research Site, Daw Park, South Australia
  - Research Site, Woodville South, South Australia
  - Research Site, Melbourne, Victoria
  - Research Site, Parkville, Victoria
  - Research Site, Nedlands, Western Australia
- Belgium (3):
  - Research Site, Jambes, Belgium
  - Research Site, Malmedy, Belgium
  - Research Site, Montigny-le-Tilleul, Belgium
- Brazil (9):
  - Research Site, Porto Alegre, Brasil
  - Research Site, Juiz de Fora, Minas Gerais
  - Research Site, Recife, Pernambuco
  - Research Site, Rio de Janeiro, Rio de Janeiro
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, Florianópolis, Santa Catarina
  - Research Site, Santo André, São Paulo
  - Research Site, São Paulo, São Paulo
  - Research Site, Rio de Janeiro
- Denmark (7):
  - Research Site, Aalborg
  - Research Site, Hellerup
  - Research Site, Hvidovre
  - Research Site, København NV
  - Research Site, Odense C
  - Research Site, Rødovre Municipality
  - Research Site, Silkeborg
- Germany (4):
  - Research Site, Berlin
  - Research Site, Erfurt
  - Research Site, Leipzig
  - Research Site, Marburg
- India (5):
  - Research Site, Hyderabad, Andhra Pradesh
  - Research Site, Bangalore, Karnataka
  - Research Site, Jaipur, Rajasthan
  - Research Site, Coimbatore
  - Research Site, Noida
- Philippines (2):
  - Research Site, Manila
  - Research Site, Quezon City
- United Kingdom (17):
  - Research Site, Dartford, Kent
  - Research Site, Hamilton, Lanarkshire
  - Research Site, Motherwell, Lanarkshire
  - Research Site, Cookstown, Northern Ireland
  - Research Site, Limavady, Northern Ireland
  - Research Site, Newtownabbey, Northern Ireland
  - Research Site, Barry, South Glamorgan
  - Research Site, Barry, Vale of Glamorgan
  - Research Site, Bradford-on-Avon, Wiltshire
  - Research Site, Airdrie
  - Research Site, Birmingham
  - Research Site, Blantyre
  - Research Site, Bolton
  - Research Site, Carrickfergus
  - Research Site, Chesterfield
  - Research Site, Coventry
  - Research Site, Hamilton

REFERENCES:
- [Derived] Partridge MR, Miravitlles M, Stahl E, Karlsson N, Svensson K, Welte T. Development and validation of the Capacity of Daily Living during the Morning questionnaire and the Global Chest Symptoms Questionnaire in COPD. Eur Respir J. 2010 Jul;36(1):96-104. doi: 10.1183/09031936.00123709. Epub 2009 Nov 6. PMID 19897551

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 706 subjects were enrolled; 264 were not randomised: 190 with eligibility not fulfilled, 11 with adverse events, 4 with discontinuation criteria, 40 voluntary discontinuations, 2 lost to follow-ups, 6 non-compliance, 1 for safety reasons, 10 with other reasons not specified. 442 subjects were randomised
Period: Period 1
Arm/Group | Symbicort Turbuhaler First, Then Seretide Diskus | Seretide Diskus First, Then Symbicort Turbuhaler
Started | 217 (This was a cross-over study) | 225
Completed | 211 | 213
Not Completed | 6 | 12
Not completed — Eligibility criteria not fulfilled | 2 | 6
Not completed — Adverse Event | 2 | 2
Not completed — Development of study-specific criteria | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Protocol Violation | 0 | 1
Period: Period 2
Arm/Group | Symbicort Turbuhaler First, Then Seretide Diskus | Seretide Diskus First, Then Symbicort Turbuhaler
Started | 211 | 213
Completed | 204 | 203
Not Completed | 7 | 10
Not completed — Adverse Event | 5 | 7
Not completed — Eligibility not fulfilled | 0 | 1
Not completed — Discontinuation criteria | 2 | 0
Not completed — Severe non-compliance | 0 | 1
Not completed — Other | 0 | 1
Period: Period 3
Arm/Group | Symbicort Turbuhaler First, Then Seretide Diskus | Seretide Diskus First, Then Symbicort Turbuhaler
Started | 204 | 203
Completed | 204 | 201
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Symbicort Turbuhaler First, Then Seretide Diskus | Seretide Diskus First, Then Symbicort Turbuhaler | Total
Number analyzed (Participants) | 217 | 225 | 442
Age Continuous [Mean (Full Range); unit: years] | 62.9 [41 to 82] | 63.2 [40 to 86] | 63.1 [40 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 71 | 126
  Male | 162 | 154 | 316

OUTCOME MEASURES:

1. Primary Outcome: Peak Expiratory Flow (PEF) 5 Minutes After Morning Dose
Description: The change from baseline in PEF was calculated using the average over baseline (the last 7 days of run-in and washout period respectively), and all days of treatment, with baseline as covariate.
Time Frame: Baseline (daily records during run-in, and washout) and daily records during the treatment period of 7 days
Population: Includes all subjects with at least one dose of study medication and who contribute sufficient data for the endpoint to be calculated.
Measure: Mean (Standard Deviation); unit: liters/minute
Groups:
- Symbicort Turbuhaler: Symbicort Turbuhaler (budesonide/formoterol) 320/9 μg
- Seretide Diskus: Seretide Diskus (salmeterol/fluticasone) 50/500 μg
Arm/Group | Symbicort Turbuhaler | Seretide Diskus
Number analyzed (Participants) | 385 | 390
liters/minute | 15.1 (28.5) | 13.4 (28.2)

2. Secondary Outcome: PEF Before Morning Dose
Description: The change from baseline was calculated using the average over baseline (the last 7 days of run-in and washout period respectively), and over all days of treatment, with baseline as covariate.
Time Frame: Baseline (daily records during run-in, and washout) and daily records during the treatment period of 7 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters/minutes
Arm/Group | Symbicort Turbuhaler | Seretide Diskus
Number analyzed (Participants) | 416 | 425
Liters/minutes | 4.8 (28.2) | 7.9 (24)

3. Secondary Outcome: PEF 15 Minutes After Morning Dose
Description: as for outcome 2
Time Frame: Baseline (daily records during run-in, and washout) and daily records during the treatment period of 7 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters/minute
Arm/Group | Symbicort Turbuhaler | Seretide Diskus
Number analyzed (Participants) | 377 | 389
Liters/minute | 19.9 (30.3) | 16.7 (28.5)

4. Secondary Outcome: PEF Before Evening Dose
Description: as for outcome 2
Time Frame: Baseline (daily records during run-in, and washout) and daily records during the treatment period of 7 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters/minute
Arm/Group | Symbicort Turbuhaler | Seretide Diskus
Number analyzed (Participants) | 418 | 426
Liters/minute | 4 (24.3) | 1.8 (50)

5. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Before Morning Dose
Description: as for outcome 2
Time Frame: Baseline (daily records during run-in, and washout) and daily records during the treatment period of 7 days
Population: Includes all subjects with at least one dose of study medication and contribute sufficient data for the endpoint to be calculated.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Symbicort Turbuhaler | Seretide Diskus
Number analyzed (Participants) | 280 | 269
Liters | 0.0310 (0.2460) | 0.0590 (0.2310)

6. Secondary Outcome: FEV1 15 Minutes After Morning Dose
Description: as for outcome 2
Time Frame: Baseline (daily records during run-in, and washout) and daily records during the treatment period of 7 days
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Symbicort Turbuhaler | Seretide Diskus
Number analyzed (Participants) | 249 | 249
Liters | 0.1220 (0.2530) | 0.1030 (0.3720)

7. Secondary Outcome: FEV1 Before Evening Dose
Description: as for outcome 2
Time Frame: Baseline (daily records during run-in, and washout) and daily records during the treatment period of 7 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Symbicort Turbuhaler | Seretide Diskus
Number analyzed (Participants) | 248 | 243
Liters | 0.1470 (0.2470) | 0.1060 (0.2010)

8. Secondary Outcome: Change in PEF From Before Dose to 5 Minutes After Dose in the Morning
Description: The change from pre-dose was calculated using the average over baseline (the last 7 days of run-in and washout period respectively), and over all days of treatment, with pre-dose run-in/washout as covariate.
Time Frame: Baseline (daily records during run-in, and washout) and daily records during the treatment period of 7 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters/minute
Arm/Group | Symbicort Turbuhaler | Seretide Diskus
Number analyzed (Participants) | 279 | 279
Liters/minute | 0.0160 (0.2) | 0.0030 (0.299)

9. Secondary Outcome: Change in PEF From Before Dose to 15 Minutes After Dose in the Morning
Description: The change from pre-dose was calculated using the average over baseline (the last 7 days of run-in and washout period respectively), and over all days of treatment, with mean pre-dose run-in/washout as covariate.
Time Frame: Baseline (daily records during run-in, and washout) and daily records during the treatment period of 7 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters/minute
Arm/Group | Symbicort Turbuhaler | Seretide Diskus
Number analyzed (Participants) | 368 | 376
Liters/minute | 11.6 (16.2) | 6.1 (16.5)

10. Secondary Outcome: Change in FEV1from Before Dose to 5 Minutes After Dose in the Morning
Description: as for outcome 9
Time Frame: Baseline (daily records during run-in, and washout) and daily records during the treatment period of 7 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Symbicort Turbuhaler | Seretide Diskus
Number analyzed (Participants) | 368 | 376
Liters | 15.8 (20.8) | 9.6 (19.9)

11. Secondary Outcome: Change in FEV1 From Before Dose to 15 Minutes After Dose in the Morning
Description: as for outcome 9
Time Frame: Baseline (daily records during run-in, and washout) and daily records during the treatment period of 7 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Symbicort Turbuhaler | Seretide Diskus
Number analyzed (Participants) | 233 | 238
Liters | 0.0930 (0.1870) | 0.0280 (0.1630)

12. Secondary Outcome: Change in FEV1 From Before Dose to 5 Minutes After Dose at the Clinic
Description: The change from pre-dose was calculated using the pre-dose baseline value (run-in and washout period respectively), and pre-dose value at day 1, with pre-dose run-in/washout as covariate.
Time Frame: Baseline (run-in, and washout) and day 1 of treatment period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Symbicort Turbuhaler | Seretide Diskus
Number analyzed (Participants) | 233 | 238
Liters | 0.1120 (0.1950) | 0.0440 (0.1640)

13. Secondary Outcome: Change in Forced Vital Capacity (FVC) From Before Dose to5 Minutes After Dose at the Clinic
Description: as for outcome 12
Time Frame: Baseline (run-in, and washout) and day 1 of treatment period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Symbicort Turbuhaler | Seretide Diskus
Number analyzed (Participants) | 415 | 426
Liters | 0.0950 (0.1370) | 0.0490 (0.1060)

14. Secondary Outcome: Capacity of Daily Living in the Morning (CDLM) (Change From Pre to End of Treatment)
Description: The change from baseline was calculated using the average over baseline (the last 7 days of run-in and washout period respectively), and over all days of treatment, with baseline as covariate. Score scale 0 - 5 with 0=worst and 5 = best.
Time Frame: Baseline (daily records during run-in, and washout) and daily records during the treatment period of 7 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Seretide Diskus First: Seretide Diskus (salmeterol/fluticasone) 50/500 μg
Arm/Group | Symbicort Turbuhaler | Seretide Diskus First
Number analyzed (Participants) | 415 | 426
units on a scale | 0.1920 (0.2530) | 0.1240 (0.2310)

15. Secondary Outcome: Difficulty in Getting Out From Bed (MASQ) (Change From Pre to End of Treatment)
Description: as for outcome 14
Time Frame: Baseline (daily records during run-in, and washout) and daily records during the treatment period of 7 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Symbicort Turbuhaler | Seretide Diskus
Number analyzed (Participants) | 319 | 311
Units on a scale | 0.21 (0.64) | 0.14 (0.75)

16. Secondary Outcome: The Clinical Chronic Obstructive Pulmonary Disease (COPD) Questionnaire (Change From Pre to End of Treatment)
Description: The change from baseline was calculated using the average over baseline (the last 7 days of run-in and washout period respectively), and over all days of treatment, with baseline as covariate. Score scale 0 - 6 with 0=worst and 6 = best.
Time Frame: Baseline (daily records during run-in, and washout) and daily records during the treatment period of 7 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Symbicort Turbuhaler | Seretide Diskus
Number analyzed (Participants) | 394 | 396
Units on a scale | 0.24 (0.75) | 0.19 (0.73)

ADVERSE EVENTS:
Arm/Group | Symbicort Turbuhaler | Seretide Diskus
Serious Adverse Events (participants affected / at risk) | 3/420 | 1/429
Other Adverse Events (participants affected / at risk) | 0/420 | 0/429
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Symbicort Turbuhaler (N=420) | Seretide Diskus (N=429)
Gait disturbance (General disorders) | 1 | 0
Chronic obstructive oulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to any publication or disclosure, the PI provides AstraZeneca with preliminary data and drafts and with the proposed final manuscript. AstraZeneca shall have a period of 30 days from receipt of the proposed final manuscript to review it and may within such time frame require that submission for publication or disclosure be delayed.